CLINICAL TRIAL: NCT07161791
Title: Exploratory Clinical Study of Camrelizumab Combined With Pirfenidone and Chemotherapy in the Treatment of Advanced Triple-Negative Breast Cancer
Brief Title: Camrelizumab, Pirfenidone, and Chemotherapy in the Treatment of Advanced Triple-Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Tong Liu, Vice President of the Affiliated Oncology Hospital of Harbin Medical University, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-271
Record Dates: First submitted 2025-08-15; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer (TNBC)
Keywords: Breast Cancer; TNBC; Immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pirfenidone; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Treatment Regimen:
  Camrelizumab: 200 mg intravenous (IV) every 3 weeks (q3w). Pirfenidone: 200 mg three times daily (tid), escalated to 600 mg tid based on tolerability.
  Chemotherapy: Investigator's choice of standard regimens (e.g., paclitaxel 175 mg/m² IV q3w or capecitabine 1000 mg/m² orally bid on days 1-14 of a 21-day cycle).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Combined With Pirfenidone and Chemotherapy Treatment Group (Experimental): Study Population:
  Patients with recurrent or metastatic triple-negative breast cancer (TNBC) who have progressed after first-line systemic therapy with immune checkpoint inhibitors (anti-PD-1/PD-L1).
  Treatment Regimen:
  Camrelizumab: 200 mg intravenous (IV) every 3 weeks (q3w). Pirfenidone: 200 mg three times daily (tid), escalated to 600 mg tid based on tolerability.
  Chemotherapy: Investigator's choice of standard regimens (e.g., paclitaxel 175 mg/m² IV q3w or capecitabine 1000 mg/m² orally bid on days 1-14 of a 21-day cycle).
  Interventions: Drug: Camrelizumab Combined With Pirfenidone and Chemotherapy

INTERVENTIONS:
Drug: Camrelizumab Combined With Pirfenidone and Chemotherapy — Treatment Regimen:
  Camrelizumab: 200 mg intravenous (IV) every 3 weeks (q3w). Pirfenidone: 200 mg three times daily (tid), escalated to 600 mg tid based on tolerability.
  Chemotherapy: Investigator's choice of standard regimens (e.g., paclitaxel 175 mg/m² IV q3w or capecitabine 1000 mg/m² orally bid on days 1-14 of a 21-day cycle).

SUMMARY:
This is a prospective, single-arm, exploratory clinical study, planned to enroll 12 patients with advanced triple-negative breast cancer who have received first-line systemic treatment with immune checkpoint inhibitors. The treatment regimen will continue until disease progression, intolerable toxicity, withdrawal of informed consent, or investigator's judgment that treatment must be terminated. Imaging assessment will be performed according to RECIST 1.1 criteria, with the research center's assessment results as the final outcome. Subjects who discontinue treatment will enter the follow-up period: 1) Safety follow-up until 30 days after the last dose; 2) Subjects who discontinue treatment for reasons other than progression disease (PD) or death will undergo efficacy follow-up until disease progression, initiation of other anti-tumor drugs, or death, whichever comes first; 3) All subjects will enter the trial period upon enrollment and receive camrelizumab combined with pirfenidone and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-70 years.
* Histologically confirmed recurrent/metastatic TNBC (ER-negative: IHC ER <1%; PR-negative: IHC PR <1%; HER2-negative: IHC -/+, or IHC ++ but FISH/CISH negative), with at least one measurable lesion per RECIST v1.1.
* ECOG performance status 0-2.
* Estimated life expectancy ≥3 months.
* Received first-line chemotherapy + PD-1/PD-L1 inhibitor for metastatic or locally advanced unresectable TNBC, with response of CR/PR or stable disease lasting ≥3 months. For neoadjuvant/adjuvant therapy, disease progression during treatment or within 6 months after completion will be considered as first-line failure.
* Adequate organ function (no transfusion, growth factor, or thrombopoietic agents within 2 weeks before screening):
* Hematology: ANC ≥1.5×10⁹/L; PLT ≥90×10⁹/L; Hb ≥90 g/L.
* Serum chemistry: TBIL ≤1.5×ULN; ALT and AST ≤1.5×ULN; ALP ≤2.5×ULN; BUN and Cr ≤1.5×ULN with creatinine clearance ≥50 mL/min (Cockcroft-Gault).
* TSH ≤ULN (if abnormal, T3 and T4 must be assessed; enrollment allowed if T3/T4 normal).
* Cardiac: LVEF ≥50% by echocardiography; 18-lead ECG with QTcF <480 ms (female).
* Women of childbearing potential must have negative pregnancy test (serum or urine) within 7 days prior to enrollment and agree to use adequate contraception during treatment and for 4 months after last dose.
* Voluntarily signed informed consent and good compliance.

Exclusion Criteria:

* Concurrent participation in another interventional cancer trial.
* Received other antitumor therapy within 14 days before first dose.
* Prior treatment with pirfenidone.
* Untreated active brain metastases or leptomeningeal disease.
* Major non-breast cancer surgery within 4 weeks prior to enrollment or incomplete recovery from such surgery.
* Active or history of autoimmune disease (except vitiligo, resolved childhood asthma without treatment in adulthood).
* Severe cardiac disease (e.g., heart failure with LVEF <50%, uncontrolled arrhythmias, angina requiring medication, significant valvular disease, recent myocardial infarction, poorly controlled hypertension >180/100 mmHg).
* Congenital or acquired immunodeficiency (e.g., HIV infection).
* Live vaccination within 4 weeks before or during study.
* Known allergy to study drugs or excipients.
* Severe concomitant disease or condition that may interfere with study participation per investigator judgment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR（Objective Response Rate） | At the end of every 2 Cycles (each cycle is 21 days) , From first treatment Cycle until achieving complete response (CR) or partialresponse (PR) per RECIST v1.1.], assessed up to 1 year.
  defined as the proportion of patients achieving complete response (CR) or partial response (PR) per RECIST v1.1.

SECONDARY OUTCOMES:
DCR（Disease Control Rate） | Patients undergo imaging evaluation in every 2 cycles（each cycyle is 21 days）until achieving SD per RECIST v1.1 or through study completion, assessed up to 1 year.
  Proportion of patients with CR, PR, or stable disease (SD) ≥6 months
CBR（Clinical Benefit Rate） | through study completion, an average of 1 year".
  Proportion of patients with CR, PR, or SD ≥6 months
PFS（Progression-Free Survival） | up to 1 year
  Time from enrollment to disease progression or death
OS（Overall Survival） | up to 1 year
  Time from enrollment to death from any cause

IPD SHARING:
Plan to Share IPD: No